CLINICAL TRIAL: NCT04227314
Title: Randomized Double Blind Controlled Trial Comparing the Safety and Efficacy of Apremilast Versus Placebo in Severe Forms of Recurrent Aphthous Stomatitis
Acronym: PREMS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019/0411/HP
Record Dates: First submitted 2019-12-13; First posted 2020-01-13 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Recurrent Aphtous Stomatitis
MeSH Terms: interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: double blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apremilast (Experimental): apremilast: 30 mg twice daily during a 12 week double blind placebo controlled period, then 30 mg twice daily during an additional 12 week active treatment period
  Interventions: Drug: Apremilast
- Placebo (Placebo Comparator): Placebo: 30 mg twice daily during the initial 12 week double blind placebo controlled period
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Apremilast — Apremilast: 30 mg twice daily during a 12 week double blind placebo controlled period, then 30 mg twice daily during an additional 12 week active treatment period
  Arms: Apremilast
Drug: Placebo oral tablet — Placebo: 30 mg twice daily during the initial 12 week double blind placebo controlled period,
  Arms: Placebo

SUMMARY:
The objective of the study is to assess the superiority of apremilast in comparison with placebo to achieve Complete Remission (CR) of oral ulcers at Week 12, in patients with severe Recurrent aphtous stomatitis resistant or intolerant to colchicine.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female patients aged ≥18 years old with severe primary RAS resistant to colchicine prescribed at a dose of 1mg/day or more for at least 3 months, or intolerant to colchicine

Severity of primary oral aphtous ulcer is defined by the presence of at least one of the following criteria:

i) - At least one giant oral ulcer (≥ 1cm in diameter) confirmed by the investigator during the month preceding inclusion and/or, ii) - Multiple simultaneous oral ulcers ( ≥4), including herpetiform ulcers confirmed by the investigator during the month preceding inclusion and/or, iii) - Continuous evolution of oral ulcers, some lesions healing, as newly appearing oral ulcers develop within the month before inclusion and/or, iv) - Oral ulcers occurring at least 7 days each month during the previous 3 months and/or v) - Major pain related to oral ulcers interfering with eating, speaking, or swallowing

- In all cases, patients must have at least one oral ulcer on the date of inclusion

2. Patient having read and understood the information letter and signed the Informed Consent Form 3. For women who are not postmenopausal and who do not plan on having children anymore: agreement to remain abstinent or use two adequate methods of contraception 4. Patient able to comply with the study protocol, in the investigator's judgment 5. Patient affiliated with, or beneficiary of a social security (health insurance) category

Exclusion Criteria:

1. Patient has any significant medical condition, significant laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
2. Patient has secondary RAS (e.g., celiac disease, Crohn's disease, ulcerative colitis, relapsing polychondritis, PFAPFA, AIDS…).
3. Depression and suicidal ideation
4. Co-medication with a cytochrome P450 3A4 (CYP3A4) enzyme inducer ( especially, rifampicin and most anti-epileptic drugs (e.g. carbamazepine, phenytoin)
5. Severely underweight patient (BMI < 18.5 kg/m2)
6. Patient cannot be followed regularly.
7. Patient has any other inflammatory oral disease, which confounds the ability to interpret data from the study (ie, lichen planus, auto immune bullous diseases with oral involvement),
8. Patient has any medical condition that requires systemic treatment which may confound the ability to interpret data from the study (ie, lupus erythematosus, rheumatoid arthritis...)
9. Patient is currently enrolled in any other therapeutic trial.
10. Other than RAS, subject has any clinically significant (as determined by the Investigator) cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic disease, or other major disease that is currently uncontrolled.
11. Malignancy or history of malignancy or myeloproliferative or lymphoproliferative disease within the past 5 years, except for treated (ie, cured) basal cell or squamous cell carcinomas, in situ cervix carcinoma, or any situation in which the oncologist in charge of the patient considers that oncologic risk allows the use of apremilast.
12. Patient with positive blood test for HIV.
13. Any bacterial infections requiring treatment with oral or injectable antibiotics, or significant viral or fungal infections, within 4 weeks of Screening. Any treatment for such infections must have been completed and the infection cured, at least 4 weeks prior to Screening and no new or recurrent infections prior to the Baseline Visit.
14. Patient has received a live vaccine within 3 months of baseline or plans to do so during study.
15. Patient is a pregnant or breastfeeding (lactating) woman or intending to become pregnant during the study; Women who are not postmenopausal (≥ 12 months of non-therapy-induced amenorrhea) or surgically sterile must have a negative result from a serum pregnancy test within 1 week prior to randomization.
16. Patient has used systemic therapy which may potentially be effective in RAS within four weeks prior to randomization (including, but not limited to corticosteroids, azathioprine, levamisole, thalidomide).
17. Patient has used biologic therapy including anti TNF within 5 pharmacokinetic half-lives.
18. Prior treatment with apremilast, or participation in a clinical study, involving apremilast.
19. Patient has any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
20. Galactose intolerance, lactase deficiency or glucose/galactose malabsorption
21. Patient is deemed unreliable or for any reason not able to comply with the protocol
22. Patient with alcohol dependency
23. Male patient intending to conceive a child with his partner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Presence of oral ulcer during clinical examination | Week 12
  Presence or absence of oral ulcer
Presence of oral ulcer during clinical examination | Week 14
  Presence or absence of oral ulcer

SECONDARY OUTCOMES:
Number of oral ulcer during clinical examination | Week 12
  Mean cumulative number of oral ulcers at the Week 12 evaluation
Number of oral ulcer during clinical examination | Week 14
  Mean cumulative number of oral ulcers at the Week 14 evaluation
Difference from baseline in quality of life | Week 14
  quality of life will be evaluated using SF36
Occurrence since baseline of severe and adverse events | Week 14
Occurrence since baseline of non-severe adverse events | Week 14

CONTACTS AND LOCATIONS:
Overall Officials: Pascal JOLY, Pr, Principal Investigator — University Hospital, Rouen

IPD SHARING:
Plan to Share IPD: No